CLINICAL TRIAL: NCT07001865
Title: Metabolically Healthy Obesity Increases the Risks of MASLD and Hyperuricemia: A Cohort Study With Mediation Analysis
Brief Title: Metabolically Healthy Obesity Increases the Risks of MASLD and Hyperuricemia
Status: Enrolling by invitation | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-073RS-01; MR-33-25-026108 (Other: medicalresearch.cn)
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolically Healthy Obesity; Hyperuricemia
MeSH Terms: conditions — Obesity, Metabolically Benign; Hyperuricemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MASLD cohort: participants with non-MASLD at baseline
- Hyperuricemia: participants with non-Hyperuricemia at baseline

SUMMARY:
Although metabolically healthy obesity (MHO) is often considered a relatively benign obesity, its association with the risk of metabolic dysfunction-associated steatotic liver disease (MASLD) and hyperuricemia remains unclear. This study examined the associations between MHO and other metabolic-obesity phenotypes with MASLD and hyperuricemia, and explored the mediating roles of metabolic indicators.This study included 11,712 and 13,846 participants from a health examination cohort at the First Affiliated Hospital of Ningbo University for MASLD and hyperuricemia analyses, respectively. Participants were classified into four metabolic-obesity phenotypes, with MHO defined as obesity without metabolic syndrome components. The outcomes were MASLD and hyperuricemia. Cox regression and mediation analyses were conducted to assess associations and mediating effects.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent comprehensive health examinations at the Physical Examination Center of the First Affiliated Hospital of Ningbo University between 2017 and 2024;
2. Aged 18 years or older at baseline;
3. Completed an abdominal ultrasound examination during the health check-up.

Exclusion Criteria:

1. Underweight status at baseline, defined as BMI < 18.5 kg/m² ；
2. Missing data on height, weight, or components of the metabolic syndrome ;
3. Baseline diagnosis of MASLD or any other liver diseases
4. Baseline diagnosis of hyperuricemia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cohort study included participants who underwent comprehensive health examinations at the Physical Examination Center of the First Affiliated Hospital of Ningbo University between 2017 and 2024. A total of 18,261 individuals aged 18 years or older who completed abdominal ultrasound examinations were initially considered. After excluding underweight individuals (BMI < 18.5 kg/m²; N = 1,138) and those with missing data on height, weight, or metabolic syndrome (MetS) components (N = 83), 17,040 participants remained eligible for further analysis.For the MASLD incidence analysis, individuals with a baseline diagnosis of MASLD or other liver diseases (N = 5,328) were excluded, resulting in 11,712 participants. For the hyperuricemia incidence analysis, those with baseline hyperuricemia (N = 3,194) were further excluded, yielding 13,846 eligible participants. During a median follow-up period of up to 7 years, 3,756 incident cases of MASLD and 3,294 incident cases of hyperuricemia were
Sampling Method: Non-Probability Sample
Enrollment: 17040 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MASLD and Hyperuricemia | 7 years
  through study completion

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University Ningbo, Zhejiang, China, 315000, Ningbo, Zhejiang Province 315000 Recruiting, Ningbo, China

IPD SHARING:
Plan to Share IPD: No